CLINICAL TRIAL: NCT00277966
Title: Cardiac Catheterization Laboratory Radiology Performance Improvement
Brief Title: Cath Lab Performance Improvement
Status: Withdrawn | Type: Observational
Why Stopped: No enrollment as this was a retrospective review, not a clinical trial.
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-051
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Congenital Disorders
Keywords: Pediatric; Cardiac Catheterization; Fluoroscopy time
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
In 2004, the Cardiac Cath Lab at Children's Healthcare of Atlanta was asked to conduct a Quality Improvement Review examining radiation exposure.

DETAILED DESCRIPTION:
In 2004, the Cardiac Cath Lab at Children's Healthcare of Atlanta was asked to conduct a Quality Improvement Review examining radiation exposure.

To perform radiological procedures with minimal radiation exposure and to ensure safe care during catheterization procedures, we conducted a chart review of all patients requiring fluoroscopy in the lab during the period of January - June, 2004.

• Based on our Retrospective Review, we were able to present Our New Standards to the Cardiac Cath Lab Committee at the end of June, 2004 with the following:

1. Diagnostic procedure time decreased from 45 minutes standard to 30 minutes standard.
2. Intervention and Electrophysiology procedure time reduced from 90 minutes to 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Medical charts of all patients requiring fluoroscopy in the cardiac catheterization lab at Children's Healthcare of Atlanta, Egleston,during January - June, 2004.

Exclusion Criteria:

* Those who did not meet inclusion criteria.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2004-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Stevens, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States